CLINICAL TRIAL: NCT00313118
Title: Determination of the Mean Values of Oxidative Stress Parameters in the Plasma of Healthy Subjects
Brief Title: Mean Values of Oxidative Stress Parameters in Healthy Subjects
Status: Withdrawn | Type: Observational
Why Stopped: Problems with recruiting
Sponsor: Selim Orguel (Other)
Collaborators: Laboratory Dr. Bayer GmbH, Stuttgart, Germany (Unknown)
Responsible Party: Sponsor-Investigator, Selim Orguel, Prof. Dr., University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 067-KOA-2005-001
Record Dates: First submitted 2006-04-10; First posted 2006-04-11 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: oxidative stress parameters

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Determination of the mean value of oxidative stress parameters in normals and of the plasma and serum levels, resp. of malondialdehyde, glutathion and superoxide dismutase in healthy subjects.

DETAILED DESCRIPTION:
In certain situations, free radicals can be generated in an exaggerated manner and can injure tissues and organs by interacting with lipids, proteins, or DNA. So, oxidative stress has been implicated in a large number of human diseases. To survive, the human body has developed a complex, efficient, and highly adaptive antioxidant defense system. The eye is also protected against oxidative stress by several mechanisms involving antioxidant enzymes such as catalase (CAT) and superoxide dismutase (SOD), as well as by low-molecular-weight antioxidants such as glutathion (GSH) and ascorbate.

Primary open-angle glaucoma (POAG) is a chronic, slowly progressive optic neuropathy, characterized by excavation of the optic nerve head (ONH) and a distinctive pattern of visual field (VF) defects. The disease is multifactorial in origin, so that besides more extensively investigated factors oxidative stress has also been proposed as a contributing factor in the etiology of glaucomatous optic neuropathy. Oxidative stress represents a harmful state defined by the presence of pathologic levels of reactive oxygen species (ROS) relative to antioxidant defense.

Therefore, it would be also important to determine whether there is a relationship between circulating levels of the defense parameters to oxidative stress like malondialdehyde, GSH and SOD, and the occurrence of POAG.

Since there are only the limits of variation for these defense parameters available, mean values of the plasma levels of malondialdehyde, glutathion and superoxide dismutase will be determined in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* German native speakers
* Age between 18-80 years
* Healthy without medication
* No ophthalmic disease

Exclusion Criteria:

* Any history of ocular or systemic diseases or of drug or alcohol abuse
* Any mentally impaired patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy persons
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-01; Primary Completion 2010-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Hospital, Basel, Switzerland
Locations (1):
- University Eye Clinic Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No